CLINICAL TRIAL: NCT01260753
Title: Double Blind Randomised Placebo and Active Controlled, Proof of Activity Study of UR-63325 in Allergic Rhinitis Induced by Nasal Challenge to Allergic Patients Otherwise Healthy
Brief Title: Proof of Activity Study of UR-63325 in Allergic Rhinitis Induced by Nasal Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palau Pharma S.L.U. (Industry)
Responsible Party: Roser Vives MD, Clinical Research Scientist, Palau Pharma S.A.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPh/00071/10; 2010-021858-20 (EudraCT Number)
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- UR-63325 (Experimental)
  Interventions: Drug: UR-63325
- Fluticasone propionate nasal spray (Active Comparator)
  Interventions: Drug: Fluticasone propionate nasal spray
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UR-63325 — UR-63325
  Arms: UR-63325
Drug: Fluticasone propionate nasal spray — Fluticasone propionate nasal spray
  Arms: Fluticasone propionate nasal spray
Drug: Placebo — Placebo to UR 63325 and fluticasone propionate nasal spray
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore the activity of UR-63325 in a model of allergic rhinitis induced by nasal allergen challenge to known allergic rhinitis patients otherwise healthy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent to participate (prior to any study-related procedures being performed) as shown by a signature on the volunteer consent form and to be able to adhere to the study restrictions and examination schedule
* Subjects with confirmed history of seasonal allergic rhinitis to grass pollen (by direct questioning of presence of positive skin prick test to pollen and History of Symptoms of allergic rhinitis) within the previous two years
* Positive skin prick test to timothy grass pollen (wheal difference with negative control ≥ 3 mm) at screening
* Subjects with positive response to screening nasal challenge with increasing doses of timothy grass pollen (Symptoms worsening with respect to the response to the diluent challenge of ≥4 points in the total nasal symptom score [TNSS]) within one hour after last nasal allergen challenge
* Screening and baseline FEV1 >80% predicted and FEV1/FVC > 70% predicted

Exclusion Criteria:

* Symptoms of allergic rhinitis within 2 weeks prior to screening
* Upper respiratory infection or sinusitis within 14 days of screening and also within 14 days of study start in each of the two periods
* Structural nasal abnormalities or nasal polyps on examination, a history of nose bleeding or recent nasal surgery
* History of asthma or asthmatic symptoms or other respiratory disease other than rhinitis within the last 2 years or FEV1<80% of predicted at screening or baseline

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Nasal and ocular symptoms scores after nasal allergen challenge | 24 hours

SECONDARY OUTCOMES:
Inflammatory parameters measured from nasal exudate | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, MD, Principal Investigator — Parexel
Locations (1):
- Parexel International GmbH, Berlin, Germany